CLINICAL TRIAL: NCT00691808
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Determine Safety and Tolerability of LX6171 Oral Suspension Dosed for 28 Days in Subjects Exhibiting Age Associated Memory Impairment (AAMI)
Brief Title: Study of LX6171 in Elderly Volunteers With Age Associated Memory Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Medical Director, Lexicon Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LX6171.1-201-AAMI; LX6171.201
Record Dates: First submitted 2008-06-02; First posted 2008-06-05 (Estimated); Results first posted 2010-03-03 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2010-02

CONDITIONS: Age-Related Memory Disorders
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Dose (Experimental)
  Interventions: Drug: LX6171 High Dose
- Low Dose (Experimental)
  Interventions: Drug: LX6171 Low Dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LX6171 High Dose — A high dose of LX6171, using an oral suspension; daily oral intake for 28 days in the morning at approximately the same time.
  Arms: High Dose
Drug: LX6171 Low Dose — A low dose of LX6171, using an oral suspension; daily oral intake for 28 days in the morning at approximately the same time.
  Arms: Low Dose
Drug: Placebo — Matching placebo dosing with daily oral intake for 28 days in the morning at approximately the same time.
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine the safety, tolerability, and effectiveness of 2 dose levels of LX6171 given over 28 days in patients with Age Associated Memory Impairment (AAMI).

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 60-80 years old.
* Complaints of memory loss in everyday life
* Non-smokers or very light smokers (no more than 10 cigarettes/day)
* Negative urine screen for drugs of abuse
* Ability to provide written informed consent

Exclusion Criteria:

* History or evidence of any disease, disorder or injury that could cause cognitive deterioration.
* Need for medications other than hormone replacement therapy, daily vitamins, or over-the-counter pain killers
* Clinically significant abnormality on electrocardiogram
* History of alcoholism or drug dependence
* Use of dietary supplements containing Huperzine A, gingko biloba, phosphatidylserine, or Docosahexaenoic acid (DHA)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip M. Brown, M.D., J.D., Study Director — Lexicon Pharmaceuticals, Inc.
Locations (2):
- Netherlands (2):
  - Kendle Netherlands, Utrecht
  - Pharmaceutical Research Associates Group BV, Zuidlaren

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed at 2 centers in the Netherlands, one in Utrecht and one in Zuidlaren. Recruitment began in October of 2007 and the last subject completed the study in October of 2008.
Groups:
- High Dose: 240 mg LX6171 oral suspension administered once per day
- Low Dose: 120 mg LX6171 oral suspension administered once per day
- Placebo: Placebo dosing volume-matched and administered once per day
Period: Overall Study
Arm/Group | High Dose | Low Dose | Placebo
Started | 35 | 36 | 32
Completed | 35 | 35 | 32
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose | Low Dose | Placebo | Total
Number analyzed (Participants) | 35 | 36 | 32 | 103
Age Continuous [Mean (Standard Deviation); unit: years] | 65.97 (3.48) | 67.81 (4.79) | 67.37 (4.41) | 67.05 (4.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 12 | 44
  Male | 19 | 20 | 20 | 59
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 0 | 1 | 1
  Black or African American | 1 | 0 | 0 | 1
  White | 34 | 36 | 31 | 101

OUTCOME MEASURES:

1. Secondary Outcome: Plasma Concentration
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | High Dose | Low Dose | Placebo
Number analyzed (Participants) | 35 | 36 | 32
ng/mL | 4670 (1470) | 2300 (618) | 0 (0)

2. Primary Outcome: Number of Participants Who Were Exposed to LX6171
Time Frame: ≥28 days
Measure: Number; unit: Participants
Arm/Group | High Dose | Low Dose | Placebo
Number analyzed (Participants) | 35 | 36 | 32
Participants | 35 | 33 | 31

3. Secondary Outcome: Change From Baseline (Day -1) in 15-Words Test: Acquisition Score at Day 28
Description: The 15-Words Test is used to measure verbal learning and memory. Subjects are scored on the number of recognized words on a scale of 0-15, with 0 being the worst and 15 being the best. The baseline (Day -1) score was subtracted from the Day 28 score to obtain the Score Change from Baseline.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: Number of words
Arm/Group | High Dose | Low Dose | Placebo
Number analyzed (Participants) | 35 | 36 | 32
Number of words | -1.2 (7.6) | -1.9 (5.6) | -1.1 (6.8)

4. Primary Outcome: Number of Participants Who Were Exposed to LX6171
Time Frame: 25 to 27 days
Measure: Number; unit: Participants
Arm/Group | High Dose | Low Dose | Placebo
Number analyzed (Participants) | 35 | 36 | 32
Participants | 0 | 2 | 1

5. Primary Outcome: Number of Participants Who Were Exposed to LX6171
Time Frame: 14 to18 days
Measure: Number; unit: Participants
Arm/Group | High Dose | Low Dose | Placebo
Number analyzed (Participants) | 35 | 36 | 32
Participants | 0 | 1 | 0

6. Secondary Outcome: Change From Baseline in 15-Word Test: Short-Term Delayed Recall Score at Day 28
Description: Subjects are asked to recall words from the preceding week's 15-Words Test. Baseline (Day -1) scores (scale 0-15, 0 being the worst) were subtracted from Day 28 scores to obtain the score change from baseline.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: Number of words
Arm/Group | High Dose | Low Dose | Placebo
Number analyzed (Participants) | 35 | 36 | 32
Number of words | -1.5 (2.3) | -1.7 (2.2) | -2.3 (2.6)

7. Secondary Outcome: Change From Baseline in Memory Assessment Clinics Self-Rating Scale Total Score at Day 28
Description: The subjects were asked to describe their memory ability in a variety of situations of everyday life (a list of 25 questions) using a 5-point scale, with a lower score being a negative assessment. Baseline (Day -1) scores were subtracted from Day 28 scores to obtain score change from baseline.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | High Dose | Low Dose | Placebo
Number analyzed (Participants) | 35 | 36 | 32
Units on a scale | 0.9 (5.9) | -2.4 (6.0) | 2.5 (6.0)

8. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index at Day 28
Description: The Pittsburgh Sleep Quality Index is a self-rated questionnaire that assesses sleep quality and disturbances. Responses were scored on a scale of 0 to 3 where 3 is the negative extreme. Baseline (Day -1) scores were subtracted from Day 28 scores to obtain score change from baseline.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | High Dose | Low Dose | Placebo
Number analyzed (Participants) | 35 | 36 | 32
Units on a scale | 0.3 (1.1) | 0.3 (1.7) | 0.7 (1.8)

9. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale at Day 28
Description: The Epworth Sleepiness Scale is a self-administered questionnaire used to help quantify a subject's level of daytime sleepiness. Subjects recorded their chances of dozing on a scale of 0 to 3, with 0 being no chance and 3 being a high chance. Baseline (Day -1) scores were subtracted from Day 28 scores to obtain score change from baseline.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | High Dose | Low Dose | Placebo
Number analyzed (Participants) | 35 | 36 | 32
Units on a scale | -0.9 (2.0) | 0 (2.6) | -0.6 (2.1)

10. Primary Outcome: Number of Subjects Reporting at Least One Adverse Event (AE)
Description: An adverse event includes any noxious, pathological, or unintended change in anatomical, physiological, or metabolic functions as indicated by physical signs or symptoms occurring in any phase of the clinical study whether or not associated with the study medication and whether or not considered related to study medication.
Time Frame: 28 days
Measure: Number; unit: Participants
Arm/Group | High Dose | Low Dose | Placebo
Number analyzed (Participants) | 35 | 36 | 32
Participants | 25 | 22 | 26

11. Primary Outcome: Number of Subjects Reporting Adverse Events Leading to Withdrawal
Time Frame: 28 days
Measure: Number; unit: Participants
Arm/Group | High Dose | Low Dose | Placebo
Number analyzed (Participants) | 35 | 36 | 32
Participants | 0 | 1 | 0

12. Primary Outcome: Treatment Compliance
Description: Subjects were considered compliant if they had taken >70% of possible doses of the study drug.
Time Frame: End of study
Measure: Mean (Standard Deviation); unit: Percentage of Participants
Arm/Group | High Dose | Low Dose | Placebo
Number analyzed (Participants) | 35 | 36 | 32
Percentage of Participants | 100.0 (0) | 99.80 (0.84) | 99.89 (0.64)

ADVERSE EVENTS:
Time Frame: 35 days
Arm/Group | High Dose | Low Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36 | 0/32
Other Adverse Events (participants affected / at risk) | 25/35 | 22/36 | 26/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose (N=35) | Low Dose (N=36) | Placebo (N=32)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 3 (3) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 7 (10)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 3 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 5 (6) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 10 (20) | 5 (8) | 9 (16)
Somnolence (Nervous system disorders) | 3 (3) | 3 (5) | 2 (2)
Early morning awakening (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Insomnia (Nervous system disorders) | 5 (5) | 2 (3) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor requires that written permission be given before the investigator can release any data publicly.